CLINICAL TRIAL: NCT05360264
Title: A Proof-of-concept, Biomarker-driven, Phase-II Clinical Trial to Explore the Activity of Decitabine Repurposing Against Advanced, Refractory, KRAS-dependent Pancreatic Ductal Adenocarcinoma (PDAC):The ORIENTATE Trial
Brief Title: tailOred dRug repurposIng of dEcitabine in KRAS-dependeNt refracTory pAncreaTic cancEr
Acronym: ORIENTATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unexpected toxicity events were documented during interim safety evaluations of the investigational drug.
Sponsor: Luca Cardone (Other)
Collaborators: Anticancer Fund, Belgium (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Catholic University of the Sacred Heart (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); San Raffaele University Hospital, Italy (Other); University of Pisa (Other)
Responsible Party: Sponsor-Investigator, Luca Cardone, Principal Investigator, Regina Elena Cancer Institute
Organization: Regina Elena Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFO21_02; 2021-002632-23 (EudraCT Number)
Record Dates: First submitted 2022-04-06; First posted 2022-05-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma Metastatic; Pancreatic Adenocarcinoma Recurrent
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental group (Experimental): A fresh, mandatory, tumor biopsy will be performed at baseline to assess KRAS mutational status and functional dependency and determine the patient's eligibility for the trial. KRAS dependency will be assessed based on computational score and inferred by a transcriptional signature of tumor cells. Transcriptomic data will be generated by using RNAseq data. Sample RNA processing and generation of the gene expression profile will be guaranteed within a maximum of 10 working days from the biopsy.
  Patients with high L-, S- or both L/S- scores of KRAS-dependency will receive DACOGEN.
  DACOGEN will be administered i.v. over 1 hour, at the dose of 10 mg/m2/d, daily on days 1-5 and 8-12 of each 4-wk cycle.
  Patients will continue to receive study treatment until objective radiological disease progression per modified RECIST 1.1, as assessed by the investigator, unacceptable toxicity, physician's decision, patient's refusal, or until they meet any other discontinuation criteria.
  Interventions: Drug: Decitabine 50 MG [Dacogen]

INTERVENTIONS:
Drug: Decitabine 50 MG [Dacogen] — DACOGEN will be administered i.v. over 1 hour, at the dose of 10 mg/m2/d, daily on days 1-5 and 8-12 of each 4-wk cycle.
  Other Names: Dacogen

SUMMARY:
The study is designed to assess the therapeutic efficacy of decitabine repurposing against advanced, refractory, ductal adenocarcinoma (PDAC) with molecular transcriptional signatures indicating dependency on the KRAS oncogene

DETAILED DESCRIPTION:
TYPE OF STUDY: Phase II study, open label, multicentre, single arm, interventional, Non-randomized ￼ TARGET POPULATION: Advanced (locally advanced or metastatic), pre-treated PDAC patients, progressing after at least one and no more than two lines of systemic therapy, whose tumors express a KRAS-dependency signature.

￼ RATIONALE. BACKGROUND: KRAS gene mutations occur in 95% of PDAC. Inhibitors targeting the prevalent KRASG12V and KRASG12D mutations in PDAC have yet to reach the clinical setting. Oncogenic KRAS-driven signatures have been derived from PDAC cancer models. Based on these, it is possible to identify a subset of PDACs that are highly addicted to oncogenic KRAS, and referred to as KRAS-dependent tumors (dKRAS), in which the direct targeting of KRAS or KRAS-dependent phenotypes reduced tumor growth. Notably, KRAS dependency was associated with a rewiring of nucleotide metabolism and the inhibition of pyrimidine biosynthesis was sufficient to inhibit the growth of dKRAS PDAC cells. In contrast, tumors that, though harboring KRAS mutations, do not display KRAS dependency are resistant to anti-KRAS targeting.

Decitabine (DEC) is FDA-approved for the treatment of myelodysplastic syndromes and acute myeloid leukaemia. Importantly, phase-I and -II clinical trials of DEC have defined a recommended phase II dose (RP2D) for DEC monotherapy in solid tumors.

HYPOTHESES AND RATIONALE: Preclinical studies show that DEC has cytotoxic activity and inhibits the growth of dKRAS PDAC, whereas KRAS-independent PDACs are not responsive. Based on solid preclinical studies and the scientific literature, the investigators' hypotheses are that: i) DEC is a potent anticancer drug inhibiting pyrimidine homeostasis and eliciting DNA damage in PDAC with a KRAS dependency; ii) The KRAS dependency of tumors can be analytically defined by computational scores based on the analysis of the gene expression signature on tumor biopsy; iii) These genetic scores might have a prognostic value. Based on these hypotheses, the investigators propose a proof-of-concept, biomarker-driven, phase-II clinical trial to explore the activity of DEC repurposing against advanced, refractory KRAS-dependent PDAC.

OBJECTIVES: The primary objective of the trial is to provide proof-of-concept of DEC antitumor activity in dKRAS metastatic PDAC.

Secondary objectives of the trial are to assess the feasibility of a molecularly tailored approach in advanced, pre-treated PDAC, as well as to assess treatment safety and tolerability, clinical benefit, impact on quality of life, and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Histologically or cytologically proven, advanced, inoperable (metastatic or locally advanced), PDAC;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2;
4. Life expectancy of at least 12 weeks;
5. At least one and no more than two lines of systemic treatment for advanced disease;
6. At least one metastatic lesion(s) and/or primary tumor amenable to pre-treatment biopsy;
7. KRAS dependency, as assessed by molecular analysis of RNA isolated from a fresh tumor biopsy;
8. Imaging-documented progressive disease (PD), according to modified RECIST 1.1 criteria;
9. Imaging-documented measurable disease, according to modified RECIST 1.1 criteria;
10. Adequate organ and marrow function;
11. Postmenopausal status or evidence of non-childbearing status (negative urine or serum pregnancy test) for women of childbearing potential;
12. Women of childbearing potential (defined as not post- menopausal for 12 months or no previous surgical sterilization) and fertile men must agree to use two highly effective forms of contraception while they are receiving

Exclusion Criteria:

1. Uncontrolled intercurrent illness(es);
2. Pregnancy or lactation;
3. Active and uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy;
4. Major surgical intervention within 4 weeks prior to enrollment;
5. Radiotherapy, surgery, chemotherapy, or an investigational therapy within 2 weeks prior to signing the treatment ICF;
6. Any previous treatment with DEC;
7. Patients with second primary cancers, except for adequately treated non- melanoma skin cancer, curatively treated in-situ cancer of the cervix, stage 1 grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) treated with curative intent and with no evidence of active disease at >1 year from the completion of curative treatment prior to study entry;
8. Persistent toxicities (≥CTCAE grade 2) caused by previous cancer therapy, excluding alopecia;
9. Serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug;
10. Serious psychiatric or medical conditions that could interfere with a valid informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Best Overall Respone (BOR) according to RECIST1.1 | From registration to date of documented best response, assessed up to 24 months
  Best response is recorded from the start of the treatment until disease progression. Tumor assessments according to modified RECIST 1.1 criteria will be performed at baseline and every 8 weeks (±1week) up to 40 weeks and then every 12 weeks (±1 week) until objective radiological disease progression according to modified RECIST criteria (evised RECIST guideline (version 1.1). Eur J Cancer 2009. DOI:10.1016/j.ejca.2008.10.026).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Every 8 weeks (±1 week) from enrolment for the first 40 weeks, then every 12 weeks (±1 week) up to discontinuation the treatment
  The percentage of patients who have achieved complete response, partial response and stable disease according to modified RECIST 1.1
Clinical Benefit Rate (CBR) | Every 8 weeks (±1 week) from enrolment for the first 40 weeks, then every 12 weeks (±1 week) up to discontinuation the treatment
  CBR is a multidimensional endpoint encompassing performance status, pain, and weight loss/gain
tumor marker (Ca19.9) response | On day 1 of every cycle and at the treatment discontinuation
  Tumor marker response is defined as percent reduction of CA19.9 at nadir, as compared to baseline levels and will be evaluated only in patients with elevated CA19.9 levels at baseline.
Number of participants with treatment-related adverse events as assessed by CTCAE version 5.0 | Adverse Events will be collected from time of signature of informed consent throughout the treatment period up to and including the 30-day follow-up period.
  Monitored throughout the study and will be assessed and graded according to CTCAE (version 5.0)
PFS (progression free survival) | Every 8 weeks (±1 week) from enrolment for the first 40 weeks, then every 12 weeks (±1 week) and at the treatment discontinuation
  PFS will be calculated form treatment start until progression or death.
OS (overall survival) | Every 8 weeks (±1 week) from enrolment for the first 40 weeks, then every 12 weeks (±1 week) and at the treatment discontinuation
  OS will be calculated from treatment start until progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: LUCA CARDONE, PhD, Principal Investigator — ISTITUTI FISIOTERAPICI OSPITALIERI- IFO - ISTITUTO REGINA ELENA; Michele Milella, Prof., Principal Investigator — AZ.OSP.UNIVERSITARIA INTEGRATA VERONA- BORGO ROMA 05091202
Locations (6):
- Italy (6):
  - Irccs S. Raffaele - Milano, Milan
  - Istituto Nazionale Tumori Di Napoli Irccs Pascale, Napoli
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Istituti Fisioterapici Ospitalieri- Ifo - Istituto Regina Elena, Rome
  - Policlinico A. Gemelli E C.I.C.- Policlinico Universitario A. Gemelli, Rome
  - Az.Osp.Universitaria Integrata Verona- Borgo Roma, Verona

IPD SHARING:
Plan to Share IPD: No